CLINICAL TRIAL: NCT00711568
Title: A Clinical Trial of Magnetic Stimulation in Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBS-014-01S; Nadeau-573-08 (Other Grant/Funding Number: University of Florida); NCT00108472 (obsolete NCT alias)
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Depression
Keywords: depression; magnetic stimulation
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Left dorsolateral frontal 20 Hz TMS delivered for 2 seconds every 30 seconds for a total of 2000 stimuli
  Interventions: Procedure: Repetitive transcranial magnetic stimulation (rTMS); Device: Repetitive Transcranial Magnetic Stimulator
- Arm 2 (Experimental): Right dorsolateral frontal 20 Hz TMS delivered for 2 seconds every 30 seconds for a total of 2000 stimuli
  Interventions: Procedure: Repetitive transcranial magnetic stimulation (rTMS); Device: Repetitive Transcranial Magnetic Stimulator
- Arm 3 (Sham Comparator): Left or right dorsolateral frontal 20 Hz sham TMS delivered for 2 seconds every 30 seconds for a total of 2000 stimuli
  Interventions: Procedure: Sham rTMS

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation (rTMS) — 20 Hz rTMS delivered for 2 seconds (40 stimuli) every 30 seconds for a total of 2000 stimuli (25 minutes)
  Arms: Arm 1; Arm 2
Procedure: Sham rTMS — 20 Hz sham rTMS delivered to L or R frontal region for 2 seconds (40 stimuli) every 30 seconds for a total of 2000 stimuli
  Arms: Arm 3
Device: Repetitive Transcranial Magnetic Stimulator — Repetitive Transcranial Magnetic Stimulator
  Arms: Arm 1; Arm 2

SUMMARY:
The purpose of this study is to determine whether repetitive high field transcranial magnetic stimulation of the left or right frontal lobes is beneficial for the treatment of depression that is refractory to antidepressant medication.

DETAILED DESCRIPTION:
Despite the utility of modern psychotropic medications, depression remains a medical problem with major societal impact. Electroconvulsive therapy (ECT) is an effective somatic treatment for depression. However, ECT has disadvantages, including risks attendant with general anesthesia and significant cognitive side effects (e.g. confusion and memory loss). An effective but safer somatic therapy for depression could help many patients.

The brain can be stimulated non-invasively by using time-varying magnetic fields to induce electrical currents within the cerebral cortex, a technique known as transcranial magnetic stimulation. Preliminary investigations have provided promising evidence of improved mood associated with high frequency repetitive transcranial magnetic stimulation (rTMS) of left prefrontal cortex in patients with medication-resistant major depression. However, the role of stimulus laterality in the effects of prefrontal rTMS have not been tested systematically. Furthermore, previous studies have likely been confounded by inadequate patient blinding and by a lack of standardization of psychotropic medication treatment. Therefore, we propose to use a carefully controlled clinical trial to directly test the hypothesis that the effects of prefrontal rTMS on mood are related to the laterality of magnetic stimulation. We also intend to improve blinding in comparison to previous studies by: 1) employing a parallel-group study design comparing real and simulated rTMS, as opposed to a crossover study design; 2) using specially constructed sham magnetic coils which can be placed directly on the scalp surface, to more effectively simulate rTMS; and 3) using trains of weak electrical impulses to simulate the cutaneous scalp stimulation associated with rTMS. We will minimize confounding effects of medications and antidepressant withdrawal by: 1) requiring that all patients have fail a monitored clinical trial of an SSRI or other comparable antidepressant prior to rTMS; and 2) continuing pharmacological treatment of depression during the rTMS phase of the trial. Demonstration of therapeutic efficacy of rTMS in this rigorously controlled clinical trial would provide a foundation for further investigation and development of this novel potential treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* All patients will meet DSM-IV criteria for Major Depressive Episode (without psychotic features).
* All patients will have a total score of 18 or higher and a score of at least 3 on item number 1 of the 24 item Hamilton Rating Scale for Depression (HAM-D).
* All patients will have failed to respond to at least two separate trials of treatment for at least 4 weeks with therapeutic dosages of antidepressant medication (including at least one SSRI) or will have been intolerant of at least three different antidepressant medications (including at least one SSRI).

Exclusion Criteria:

* Patient medications will be reviewed prior to enrollment in this study. Patients taking medications that may lower seizure threshold (e.g. metronidazole) will be excluded if the particular medication cannot be stopped or altered without affecting the patient's routine medical care.
* History of neurological illness, epilepsy or seizure disorder, intracranial tumor, or major head trauma leading to loss of consciousness of any length.
* Evidence of central nervous system disease based on baseline complete neurological examination, EEG and contrast-enhanced computerized tomography or magnetic resonance imaging of the brain.
* History of implanted pacemaker or medication pump, metal plate in skull, or metal objects in the eye or skull.
* Axis II diagnosis of Cluster A (paranoid, schizoid, or schizotypal) or Cluster B (antisocial, borderline, histrionic, or narcissistic) personality disorder.
* Axis II diagnosis of mental retardation.
* History of schizophrenia, schizoaffective disorder, other functional psychosis, rapid-cycling bipolar illness, or alcohol or drug abuse within the past year.
* Need for rapid clinical response due to conditions such as inanition, psychosis, or suicidality (defined as suicide attempt during the current major depressive episode or having a specific plan for committing suicide).
* A medical condition that is not well controlled, such as diabetes or hypertension, or concomitant medical or nutritional problems necessitating hospitalization.
* Patients taking anticonvulsant mood stabilizers (e.g. carbamazepine, valproic acid).
* Patients otherwise unable to grant informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-10; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale | Baseline x 2, end of treatment, one week, one month and 3 months post-treatment

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline x 2, end of treatment, one week, one month and 3 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E. Nadeau, MD BS BS, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

REFERENCES:
- [Background] Triggs WJ, McCoy KJ, Greer R, Rossi F, Bowers D, Kortenkamp S, Nadeau SE, Heilman KM, Goodman WK. Effects of left frontal transcranial magnetic stimulation on depressed mood, cognition, and corticomotor threshold. Biol Psychiatry. 1999 Jun 1;45(11):1440-6. doi: 10.1016/s0006-3223(99)00031-1. PMID 10356626
- [Derived] Nadeau SE, Bowers D, Jones TL, Wu SS, Triggs WJ, Heilman KM. Cognitive effects of treatment of depression with repetitive transcranial magnetic stimulation. Cogn Behav Neurol. 2014 Jun;27(2):77-87. doi: 10.1097/WNN.0000000000000031. PMID 24968008
- [Derived] Nadeau SE, Davis SE, Wu SS, Dai Y, Richards LG. A pilot randomized controlled trial of D-cycloserine and distributed practice as adjuvants to constraint-induced movement therapy after stroke. Neurorehabil Neural Repair. 2014 Nov-Dec;28(9):885-95. doi: 10.1177/1545968314532032. Epub 2014 Apr 26. PMID 24769437
- [Derived] Triggs WJ, Ricciuti N, Ward HE, Cheng J, Bowers D, Goodman WK, Kluger BM, Nadeau SE. Right and left dorsolateral pre-frontal rTMS treatment of refractory depression: a randomized, sham-controlled trial. Psychiatry Res. 2010 Aug 15;178(3):467-74. doi: 10.1016/j.psychres.2010.05.009. Epub 2010 Jun 18. PMID 20643486